CLINICAL TRIAL: NCT02823197
Title: An Intervention to Promote Active Transport for Short Distance Travel in Older Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2011/288
Record Dates: First submitted 2016-05-10; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-06

CONDITIONS: Transport Behaviour Intervention
Keywords: determinants; active transport; intervention; adolescents

ARMS (3):
- active transport lesson (Experimental): Participants receive a 2-hour lesson (at school) promoting active transport for short distance travel to various destinations.
  Interventions: Other: Active transport lesson
- active transport lesson and Facebook group (Experimental): Participants receive a 2-hour lesson (at school) promoting active transport for short distance travel to various destinations. Furthermore, they are asked to join a Facebook group on active transport in which 3 messages per week are posted during an eight-week period. The Facebook posts aim to promote the use of active transport for short distance travel.
  Interventions: Other: Active transport lesson and Facebook group
- control group (No Intervention): Participants in the control group do not receive the active transport lesson or the Facebook group.

INTERVENTIONS:
Other: Active transport lesson
  Arms: active transport lesson
Other: Active transport lesson and Facebook group
  Arms: active transport lesson and Facebook group

SUMMARY:
The purpose of this study is to determine whether a theory- and evidence-based intervention aiming to promote active transport for short distance travel among older adolescents is effective in increasing attitude, subjective norm, self-efficacy, awareness and habit towards active transport, and intention to use active transport after obtaining a driving license.

ELIGIBILITY:
Inclusion Criteria:

* must understand Dutch
* must participate in the project 'Driving License at School' of the Flemish Foundation for Traffic Knowledge

Exclusion Criteria:

* being younger than 16 years old or older than 19 years old
* already having a driving license

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 860 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in perceived benefits towards active transport | The outcome will be measured at baseline (before start intervention), posttest (1 week after the intervention) and follow-up (8 weeks after the intervention)
  Perceived benefits towards active transport (e.g. health, cost, parking lot, independence,...) will be assessed via seventeen items with a five-point answer format.
Change in perceived barriers towards active transport | The outcome will be measured at baseline (before start intervention), posttest (1 week after the intervention) and follow-up (8 weeks after the intervention)
  Perceived barriers towards active transport (e.g. time, accidents, weather, sweating,...) will be assessed via twenty-one items with a five-point answer format.
Change in subjective norm towards active transport | The outcome will be measured at baseline (before start intervention), posttest (1 week after the intervention) and follow-up (8 weeks after the intervention)
  Subjective norm towards active transport will be assessed via three items (family, friends, partner) with a five-point answer format.
Change in self-efficacy towards active transport | The outcome will be measured at baseline (before start intervention), posttest (1 week after the intervention) and follow-up (8 weeks after the intervention)
  Self-efficacy towards active transport (e.g. bad weather, darkness, when tired,...) will be assessed via eleven items with a five-point answer format.
Change in awareness towards active transport | The outcome will be measured at baseline (before start intervention), posttest (1 week after the intervention) and follow-up (8 weeks after the intervention)
  Awareness towards active transport (e.g. ecology, health benefits, private car ownership,...) will be assessed via eight items with a five-point answer format.
Change in habit towards active transport | The outcome will be measured at baseline (before start intervention), posttest (1 week after the intervention) and follow-up (8 weeks after the intervention)
  Habit towards active transport (e.g. walking or cycling for transport is something I automatically do) will be assessed via four items with a five-point answer format.
Change in intention to use active transport after obtaining a driving license | The outcome will be measured at baseline (before start intervention), posttest (1 week after the intervention) and follow-up (8 weeks after the intervention)
  Intention to use active transport after obtaining a driving license will be assessed via three items with a five-point answer format (e.g. how much do you want to keep using active transport for short distances after obtaining a driving licence).